CLINICAL TRIAL: NCT05931016
Title: Impact of Surgical Mask, FFP2 (Filtering Face Piece Class 2) Mask and FFP3 (Filtering Face Piece Class 3) Mask (With and Without Exhalation Valve) on Exercise Tolerance and Blood Gas Parameters of Patients With Known Lung Disease and Long-term Oxygen Therapy
Brief Title: Impact of Surgical Mask, FFP2 Mask and FFP3 Mask (With and Without Exhalation Valve) on Exercise Tolerance and Blood Gas Parameters of Patients With Known Lung Disease and Long-term Oxygen Therapy
Acronym: FFP-O2
Status: Completed | Type: Observational
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Maximilian Malfertheiner, PD Dr. Maximilian Malfertheiner, University Hospital Regensburg
Other Study IDs: 22-3165-101
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Face Mask; Longterm Oxygen Therapy
MeSH Terms: interventions — Walk Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with known lung disease and LTOT (long term oxygen therapy): Patients with i.e. interstitial lung, emphysema, pulmonary hypertension or COPD with the need for LTOT
  Interventions: Diagnostic Test: 6-MWT; Diagnostic Test: Spiroergometry

INTERVENTIONS:
Diagnostic Test: 6-MWT — Measurement of saturation and blood gas parameters under 6-MWT with different masks.
  Other Names: Six minutes walk test
Diagnostic Test: Spiroergometry — Measurement of saturation and blood gas parameters under spiroergometry with different masks.

SUMMARY:
The aim of the study is to find out how blood gas parameters change under the use of surgical mask, FFP2 masks and FFP3 masks (with and without exhalation valve) in patients with known lung disease and long-term oxygen therapy.

In particular, the question arises whether patients become hypoxemic or hypercapnic by using a mask. Or whether wearing a mask increases oxygen saturation by its reservoir function.

ELIGIBILITY:
Inclusion Criteria:

* Known lung disease and
* LTOT
* informed consent

Exclusion Criteria:

* Severe disease with contraindication for stress testing (e.g. myocardial infarction, acute pulmonary embolism, acute heart failure)
* Acute exacerbation of lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known lung disease hospitalized at normal wards.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Increase in capillary oxygen partial pressure | At the end of 6-MWT or spiroergometry
Increase in capillary carbon dioxide partial pressure | At the end of 6-MWT or spiroergometry

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Donaustauf, Donaustauf, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No